CLINICAL TRIAL: NCT03572803
Title: Comparative Research Among 3 Action Protocol in Other to Approach Chronic Lateral Epicondyle Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad San Jorge (Other)
Collaborators: University of Seville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C3P_CLET
Record Dates: First submitted 2018-06-14; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-03

CONDITIONS: Tendinopathy
Keywords: ntratissue Percutaneous Electrolysis; Dry needling; Eccentric exercise; Lateral epicondyle
MeSH Terms: conditions — Tendinopathy | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group of Dry Needling (Active Comparator): They will receive a treatment of dry needling, guided by ultrasound, together with a self-treatment program at home based on eccentric exercises and stretching.
  The needle will get in the relevant zone of treatment. The punction will be realized using Hong's technique (fast in-out). Three needle insertions will be carried out in the target area during 3 seconds
  Interventions: Other: Group of Dry Needling
- Group of electrolysis (Active Comparator): They will receive a treatment of Intratissue Percutaneous Electrolysis, guided by ultrasound, together with a self-treatment program at home based on eccentric exercises and stretching.
  The needle will get in the relevant zone of treatment. The punction will be realized simulating Hong's technique (fast in-out). Three needle insertions will be carried out in the target area during 3 seconds and 3mA each one.
  Interventions: Other: Group of Electrolysis
- Control Group (Sham Comparator): They will receive a treatment of punction sham, guided by ultrasound, together with a self-treatment program at home based on eccentric exercises and stretching.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Group of Dry Needling — Every group will receive a total of 3 treatment sessions distributed throughout 4 weeks of treatment. The program of eccentric exercises will be done by participants at home 5 days a week, two times a day.
  Arms: Group of Dry Needling
Other: Group of Electrolysis — Every group will receive a total of 3 treatment sessions distributed throughout 4 weeks of treatment. The program of eccentric exercises will be done by participants at home 5 days a week, two times a day.
  Arms: Group of electrolysis
Other: Control Group — Every group will receive a total of 3 treatment sessions distributed throughout 4 weeks of treatment. The program of eccentric exercises will be done by participants at home 5 days a week, two times a day.
  Arms: Control Group

SUMMARY:
The accomplishment of a treatment with Intratissue Percutaneous Electrolysis of additional form to the accomplishment of eccentric exercises and stretching program in patients with chronic lateral epicondyle tendinopathy is more effective than the accomplishment of an additional treatment with dry needling or eccentric exercises program realized of isolated form.

DETAILED DESCRIPTION:
Experimental study randomized with double blind, whose purpose is to compare three protocols in those who apply different protocols of physical therapy to themselves in three groups of intervention with patients with chronic lateral epicondyle tendinopathy.

There take part in this study people of both sexes, with ages between 18 and 65 years, all of them present chronic lateral epicondyle tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Patients diagnosed of chronic lateral epicondyle tendinopathy with a minimum of 3 months of evolution.
* Pain when palpating the lateral epicondyle area.
* Positive test in at least 1 of the following 3 clinical tests: Cozen, Thomson or Mill's
* Have the capacity to perform all clinical tests, understand the study process, and obtain informed consent.

Exclusion Criteria:

* Previous history of direct trauma, fractures, joint instability, surgery or rheumatic alterations of the lateral epicondyle area.
* Full elbow extension limited.
* Alterations at cervical level such as: cervical radiculopathy (C4-C7), degenerative pathology in the cervical spine, exacerbated pain increase with neck movements or cervical compression.
* Symptoms compatible with entrapment of the posterior interosseous nerve.
* NSAID intake the week before the intervention;
* Have received treatment with infiltration in the last year;
* Have received physiotherapy treatment during the last month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in quality of life by DASH | Pre-intervention; Post-intervention (1 week after); Follow up (26 and 52 weeks after)
  The Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure is a 30-item, self-report questionnaire designed to help describe the disability experienced by people with upper-limb disorders and also to monitor changes in symptoms and function over time. The DASH Outcome Measure contains one optional, four-item modules intended to measure symptoms and function in workers whose jobs require a high degree of physical performance.

SECONDARY OUTCOMES:
Pain, as measured by Visual Analog Scale | Pre-intervention; Intervention (4 weeks); Post-intervention (1 week after), Follow up (26 and 52 weeks after)
  Participants will be explained that a score of 0 indicates the absence of pain whereas a score of 10 represents the maximum tolerable pain.
Pressure pain thresholds (PPTs) | Pre-intervention; Intervention (4 weeks); Post-intervention (1 week after), Follow up (26 and 52 weeks after)
  Level of pressure tolerated by the patient just before feeling pain. The pressure is done with a digital algometer Type II(Somedic). PPTS will be assessed bilaterally in extensor carpi radialis brevis tendon and tibialis anterior muscle.
Pain free grip strength | Pre-intervention; Intervention (4 weeks); Post-intervention (1 week after), Follow up (26 and 52 weeks after)
  Grip strength before feeling pain. The tool used is a hydraulic hand dynamometer (Baseline). Subjects will be asked to gradually increase the grip strength while the elbow is extended and pronated and arm alongside of the body. They will be asked to stop when pain is felt. We will take three measures with each elbow.
Thickness of the tendon, as measured by ultrasound scan | Pre-intervention; Post-intervention (1 week after); Follow up (26 and 52 weeks after)
  Tendon structure
Hypervascularity, as measured by ultrasound scan | Pre-intervention; Post-intervention (1 week after); Follow up (26 and 52 weeks after)
  Tendon structure

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mª Galán Díaz, MD, Principal Investigator — Universidad San Jorge; Pablo Herrero Gallego, PhD, Study Director — Universidad San Jorge; Cleofas Rodríguez Blanco, PhD, Study Director — University of Seville
Locations (1):
- Opel España, Figueruelas, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Undecided